CLINICAL TRIAL: NCT03139591
Title: Comparison Between Lidocaine Inhalation and Intravenous Dexamethasone to Reduce Pain After Laryngeal Mask Insertion
Brief Title: Comparison Between Lidocaine Inhalation and Intravenous Dexamethasone in Reducing Pain After Laryngeal Mask Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Susilo Chandra, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes014
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Adult Patients Undergoing Elective Surgery With General Anesthesia and LMA Insertion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine inhalation (Active Comparator): Lidocaine inhalation group: 1.5 mg/kg body weight (BW) of 2% lidocaine inhalation, diluted with 2-3 ml of normal saline until the total volume was 6 ml, and intravenous normal saline injection
  Interventions: Drug: lidocaine inhalation; intravenous dexamethasone
- intravenous dexamethasone (Active Comparator): Intravenous dexamethasone group: normal saline inhalation and 10 mg of intravenous dexamethasone
  Interventions: Drug: lidocaine inhalation; intravenous dexamethasone

INTERVENTIONS:
Drug: lidocaine inhalation; intravenous dexamethasone — 1.5 mg/kg body weight (BW) of 2% lidocaine inhalation, diluted with 2-3 ml of normal saline until the total volume was 6 ml, and intravenous normal saline injection; Intravenous dexamethasone group: normal saline inhalation and 10 mg of intravenous dexamethasone.

SUMMARY:
This study aimed to compare the efficacy between lidocaine inhalation vs intravenous dexamethasone to reduce pain after laryngeal mask insertion

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups (Lidocaine inhalation and Intravenous dexamethasone group). Intravenous (IV) cannula (18 or 20 G) , non-invasive blood pressure monitor, and pulse-oxymetry had been set on the subjects 10 minutes before anesthesia began. Vital signs were recorded. Lidocaine group received 1.5 mg/kg body weight (BW) of 2% lidocaine inhalation, diluted with 2-3 ml of normal saline until the total volume was 6 ml, and intravenous normal saline injection. Dexamethasone group received normal saline inhalation and 10 mg of intravenous dexamethasone. Subjects, authors, or inhalation giver were not aware of the content of any drug given. Coinduction was done using 0.05mg/kg BW of midazolam and 2mcg/kg BW of fentanyl 5 minutes before the laryngeal mask airway (LMA) insertion. Induction was done using 2 mg/kg BW of 1% propofol and 0.5 mg/kg BW of atracurium 3 minutes before LMA insertion. Subjects were then given oxygenation using face mask without oropharyngeal airway. LMA was lubricated with normal saline. After 3 minutes of oxygenation, LMA was inserted using standard method. The LMA cuff was inflated with cuff pressure gauge of approximately 40 mmHg. After the position of LMA was confirmed to be correct, fixation was done using a tape. Maintenance of anesthesia was done using 50% oxygen in compressed air, 1% isoflurane, and atracurium. Thirty minutes before the surgery ended, 1 gram of paracetamol was given in 15 minutes as post-surgery analgetic. After the surgery was ended, subjects were given 0.04 mg/kg BW of neostigmine and 0.02 mg/kg BW of atropine. Mucus suction was performed on oropharynx and oral cavity gently, by using suction catheter 12F when subjects were still under anesthesia. After spontaneous breaths occured, LMA cuff was deflated and LMA was removed. Ventilation was continued using face mask without oropharyngeal airway. At the recovery room, pain on throat was assessed using Numerical Rating Scale. Assessment was done 2 hours after surgery in the recovery room after subjects were fully alert with Aldrette score of 10. Throat pain was assessed during rest or swallowing. In addition, subjects were asked whether or not they experienced difficulty in swallowing or hoarseness.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 20-59 years old, with American Society of Anesthesiologists (ASA) physical status of I-II who were planned to undergo any elective surgery at operating room in general anesthesia and needed LMA insertion
* Mallampati class I or II
* subjects had been explained about the study, and agreed to enroll and have signed the informed consent form
* Subjects without history of throat pain

Exclusion Criteria:

* Subjects with cardiovascular disease, history of analgetic and steroid before surgery, surgical site of neck, oral cavity, pharynx, and larynx
* Subjects with upper respiratory tract infection
* Subjects with history of drug allergy used in the trial and possibility of difficult airway
* Pregnant, obese, active smoking, uncontrolled diabetic and hypertension subjects
* Subjects with history of peptic ulcer disease.

Dropout Criteria:

* Subjects whose LMA insertion attempts more than once
* Subjects with surgery duration > 150 minutes
* Subjects who needed mechanical ventilation after surgery, subjects who vomitted
* Subjects whose LMA converted to endotracheal tube during surgery
* Subjects who received additional opioid during surgery

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | Day 1
  Numerical rating scale for throat pain

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] An J, Shin SK, Kim KJ. Laryngeal mask airway insertion in adults: comparison between fully deflated and partially inflated technique. Yonsei Med J. 2013 May 1;54(3):747-51. doi: 10.3349/ymj.2013.54.3.747. PMID 23549825
- [Background] Seet E, Yousaf F, Gupta S, Subramanyam R, Wong DT, Chung F. Use of manometry for laryngeal mask airway reduces postoperative pharyngolaryngeal adverse events: a prospective, randomized trial. Anesthesiology. 2010 Mar;112(3):652-7. doi: 10.1097/ALN.0b013e3181cf4346. PMID 20179502
- [Background] Uzture N, Menda F, Bilgen S, Keskin O, Temur S, Koner O. The Effect of Flurbiprofen on Postoperative Sore Throat and Hoarseness After LMA-ProSeal Insertion: A Randomised, Clinical Trial. Turk J Anaesthesiol Reanim. 2014 Jun;42(3):123-7. doi: 10.5152/TJAR.2014.35693. Epub 2014 Mar 11. PMID 27366405
- [Background] Sun L, Guo R, Sun L. Dexamethasone for preventing postoperative sore throat: a meta-analysis of randomized controlled trials. Ir J Med Sci. 2014 Dec;183(4):593-600. doi: 10.1007/s11845-013-1057-0. Epub 2013 Dec 20. PMID 24357270
- Available data/document: Textbook — https://books.google.co.id/books/about/Laryngeal_Mask_Anesthesia.html?id=XBJsAAAAMAAJ&redir_esc=y — Problems. In: Brimacombe JR. Laryngeal Mask Anesthesia principles and practice. London: Saunders Ltd, 2004;551-71.